CLINICAL TRIAL: NCT04038047
Title: A Prospective Study to Evaluate Biological and Clinical Effects of Significantly Corrected CFTR Function (The PROMISE Study)
Brief Title: A Prospective Study to Evaluate Biological and Clinical Effects of Significantly Corrected CFTR Function
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Nicole Hamblett (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor of Pediatrics, Division of Pulmonary and Sleep Medicine, University of Washington School of Medicine Adjunct Professor, Biostatistics, University of Washington School of Medicine Co-Executive Director, Cystic Fibrosis Therapeutics Development, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: PROMISE-OB-18
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
Keywords: CF; CFTR modulator; triple combination therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Core: Serum, Plasma, Buffy Coat, Urine, Optional Human Nasal Epithelial (cell) (HNE) Airway: Sputum GI Health: Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Core: Cystic Fibrosis patients prescribed elexacaftor, tezacaftor and ivacaftor CFTR modulator therapy (TCT).

SUMMARY:
This is a prospective, multi-center observational study. The study is designed to measure the clinical effectiveness of elexacaftor, tezacaftor and ivacaftor (ETI) triple combination therapy in people with one or more copies of the F508del mutation, study the effects of ETI across a number of CF disease manifestations, and collect specimens for future research. Subjects in the study will have one "before TCT" visit within 30 days before initiation of the therapy and five "after TCT" visits over a 30-month follow-up period. Participants who have participated in the original PROMISE cohort have the option of participating in a long-term extension with annual visits performed at the 42- and 54-month timepoints. The durability of the clinical and biological changes in PROMISE can be assessed with extended follow-up, which would enable the sub-studies to consider potential clinical consequences of the biological or physiological effects being studied. This work will help to inform long term prognosis and feasibility of certain clinical trials outcomes for interventional studies and may be useful when considering research priorities in drug development. Most participating sites have been divided into sub-study groups; each sub-study group has specific non-optional procedures conducted in addition to the "Core" procedures. Finally, there is one optional procedure (transient elastography) that will be offered to subjects at certain sites. The duration of participation for each subject is 30 months (with an additional 24 months if participants agree to the optional long-term extension). NOTE: FDA has reviewed the New Drug Application (NDA) for elexacaftor, tezacaftor and ivacaftor and has granted approval.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive genetic disorder caused by mutations in the gene encoding the cystic fibrosis transmembrane conductance regulator (CFTR) protein. In people with CF, this manifests as dysfunction in multiple organ systems including the lungs, pancreas, liver, intestines, skin and others.

While nearly 2000 mutations have been described, the most common disease-causing CFTR mutation is F508del, which is found in >85% of patients followed in the US CF Patient Registry. Two CFTR corrector drugs plus the potentiator ivacaftor have been developed as a triple combination therapy for CF patients with one or two copies of the F508del mutation. We predict that over 90% of CF patients (initially age 12 y/o and above) will be eligible for highly effective CFTR modulator therapy in the U.S.

The PROMISE study is designed to measure the direct and indirect CFTR-dependent anion secretion by collecting and analyzing clinical research outcomes and biomarkers on a large number of patients both before and after they begin treatment with elexacaftor, tezacaftor and ivacaftor triple combination therapy (TCT). This study will investigate the impact of TCT across a wide range of CF disease manifestations and organ systems. While specific biomarkers of special interest have been selected for detailed analysis in this study, an additional important goal is to collect blood, urine, stool, and airway epithelial cell specimens for long-term storage in a biorepository to enable future research. These samples can be made available for research beyond the current scope of work. The PROMISE study will provide a coordinated collection of clinical research outcomes data that can be linked with these specimens.

ELIGIBILITY:
Inclusion Criteria:

1. All genders within the age limit of the FDA approved indication for elexacaftor, tezacaftor and ivacaftor triple combination therapy (TCT) at Day 1.
2. Diagnosis of CF.
3. CFTR mutations consistent with the FDA approved indication for elexacaftor, tezacaftor and ivacaftor triple combination therapy (TCT).
4. Physician intent to prescribe elexacaftor, tezacaftor and ivacaftor triple combination therapy (TCT).
5. Willing to fast for 8 hours prior to all study visits (for subjects on overnight enteric tube feedings, willing to hold the feeding for at least 8 hours).
6. Able to perform the testing and procedures required for this study, as judged by the investigator.
7. Enrolled in the Cystic Fibrosis Foundation Patient Registry.
8. Clinically stable with no significant changes in health status within the 14 days prior to Visit 1.

Exclusion Criteria:

1. Use of any TCT within the 180 days prior to Visit 1.
2. Any acute use of antibiotics (oral, inhaled or IV) or systemic corticosteroids within the 2 weeks prior to Visit 1 for lower respiratory tract symptoms.
3. Initiation of any new chronic therapy (e.g., ibuprofen, Pulmozyme®, hypertonic saline, azithromycin, inhaled tobramycin, Cayston®, Kalydeco, Orkambi®, Symdeko®) within the 4 weeks prior to Visit 1.
4. Use of an investigational agent within the 28 days prior to Visit 1.
5. Use of chronic oral corticosteroids (equivalent to 10 mg. or more per day of prednisone) within the 28 days prior to Visit 1.
6. Treatment for nontuberculous mycobacterial (NTM) infection, consisting of ≥ two antibiotics (oral, IV, and/or inhaled) within the 28 days prior to Visit 1.
7. History of lung or liver transplantation, or listing for organ transplantation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Cystic Fibrosis, prescribed the elexacaftor, tezacaftor and ivacaftor CFTR modulator therapy (TCT).
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Sweat Chloride at 6 months | 6 months
  Change in sweat chloride from Baseline to 6 months.
Sweat Chloride at 30 months | 30 months
  Change sweat chloride from Baseline to 30 months.
Forced expiratory volume at one second (FEV1) at 6 months | 6 months
  Change in FEV1 from Baseline to 6 months.
Forced expiratory volume at one second (FEV1) at 30 months | 30 months
  Change in FEV1 from Baseline to 30 months.

SECONDARY OUTCOMES:
Weight at 6 Months | 6 months
  Change in weight from Baseline to 6 months.
Weight at 30 Months | 30 months
  Change in weight from Baseline to 30 months.
BMI at 6 Months | 6 months
  Change in BMI from Baseline to 6 months.
BMI at 30 months | 30 months
  Change in BMI from Baseline to 30 months.
Cystic Fibrosis Questionnaire Revised (CFQ-R) at 6 Months | 6 months
  Change in CFQ-R (respiratory domain) from Baseline to 6 months.
Cystic Fibrosis Questionnaire Revised (CFQ-R) at 30 months | 30 months
  Change in CFQ-R (respiratory domain) from Baseline to 30 months.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rowe, MD, Principal Investigator — University of Alabama at Birmingham; David Nichols, MD, Principal Investigator — University of Washington
Locations (56):
- United States (56):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta and Emory University, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University Harper University Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Cystic Fibrosis Center of Western New York, Buffalo, New York
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - Northwell CF Center, New York, New York
  - Children's Hospital of New York, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center/Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Cystic Fibrosis Program, Cleveland, Ohio
  - Oklahoma Cystic Fibrosis Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Cystic Fibrosis Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagel SD, Poore TS, Wagner BD, Xie J, Heltshe SL, Cross M, Bratcher PE, Taylor-Cousar JL, Wilson A, McBennett K, Morgan SJ, Singh PK, Nichols DP, Kelly A, Solomon GM. Long-term Reductions in Inflammation in People with Cystic Fibrosis Treated with Elexacaftor/Tezacaftor/Ivacaftor. Ann Am Thorac Soc. 2025 Sep 17:10.1513/AnnalsATS.202507-817OC. doi: 10.1513/AnnalsATS.202507-817OC. Online ahead of print. PMID 40961158
- [Derived] Pittman JE, Morgan S, McCreary M, Vu PT, Jorth P, Heltshe S, Hoffman LR, Kelly A, Sagel SD, Singh PK, Solomon GM, Rosenfeld M, Ratjen F; PROMISE Pediatric substudy Investigators. Clinical Effectiveness of Elexacaftor/Tezacaftor/Ivacaftor in 6- to 11-Year-Olds with Cystic Fibrosis: An Observational Study. Ann Am Thorac Soc. 2025 Nov;22(11):1696-1708. doi: 10.1513/AnnalsATS.202501-103OC. PMID 40540670
- [Derived] Nichols DP, Morgan SJ, Skalland M, Vo AT, Van Dalfsen JM, Singh SB, Ni W, Hoffman LR, McGeer K, Heltshe SL, Clancy JP, Rowe SM, Jorth P, Singh PK; PROMISE-Micro Study Group. Pharmacologic improvement of CFTR function rapidly decreases sputum pathogen density, but lung infections generally persist. J Clin Invest. 2023 May 15;133(10):e167957. doi: 10.1172/JCI167957. PMID 36976651
- [Derived] Schwarzenberg SJ, Vu PT, Skalland M, Hoffman LR, Pope C, Gelfond D, Narkewicz MR, Nichols DP, Heltshe SL, Donaldson SH, Frederick CA, Kelly A, Pittman JE, Ratjen F, Rosenfeld M, Sagel SD, Solomon GM, Stalvey MS, Clancy JP, Rowe SM, Freedman SD; Promise Study Group. Elexacaftor/tezacaftor/ivacaftor and gastrointestinal outcomes in cystic fibrosis: Report of promise-GI. J Cyst Fibros. 2023 Mar;22(2):282-289. doi: 10.1016/j.jcf.2022.10.003. Epub 2022 Oct 21. PMID 36280527
- [Derived] Nichols DP, Paynter AC, Heltshe SL, Donaldson SH, Frederick CA, Freedman SD, Gelfond D, Hoffman LR, Kelly A, Narkewicz MR, Pittman JE, Ratjen F, Rosenfeld M, Sagel SD, Schwarzenberg SJ, Singh PK, Solomon GM, Stalvey MS, Clancy JP, Kirby S, Van Dalfsen JM, Kloster MH, Rowe SM; PROMISE Study group. Clinical Effectiveness of Elexacaftor/Tezacaftor/Ivacaftor in People with Cystic Fibrosis: A Clinical Trial. Am J Respir Crit Care Med. 2022 Mar 1;205(5):529-539. doi: 10.1164/rccm.202108-1986OC. PMID 34784492